CLINICAL TRIAL: NCT06670560
Title: Onco-Respirology Epidemiology Based on Real-world Big Data in Respiratory Medicine
Status: Active, not recruiting | Type: Observational
Sponsor: Zhou Chengzhi (Other)
Responsible Party: Sponsor-Investigator, Zhou Chengzhi, Clinical Professor, Guangzhou Institute of Respiratory Disease
Organization: Guangzhou Institute of Respiratory Disease (Other)
Other Study IDs: CROC-24-10
Record Dates: First submitted 2024-10-31; First posted 2024-11-01 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Respiratory; Epidemiology; Neoplasms
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this observational study is to understand the changes in the types of respiratory patients hospitalized in China in recent years through a multicenter retrospective clinical study, and at the same time to understand the reasons for hospitalization and the distribution of different tumor types in oncology patients, so as to provide data support and theoretical basis for the future development of China's respiratory department.

The main questions it aims to answer are

1. the trend of change of respiratory diseases in China in the past 10 years.
2. the trend of change in the causes of hospitalization of respiratory tumor patients in China in the past 10 years.
3. the trend of the proportion of each tumor in the respiratory department in China over the past 10 years.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of Respiratory diseases Must be an inpatient

Exclusion Criteria:

Non-respiratory inpatients

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A respiratory oncology epidemiology study based on real-world big data from respiratory medicine, with retrospective data collected from respiratory medicine inpatients at a multicenter for nearly 10 years.
Sampling Method: Non-Probability Sample
Enrollment: 100000 (Estimated)
Dates: Start 2024-09-05 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
proportion | 10 years
  1. to explore the trend of respiratory diseases (COPD, asthma, bronchiectasis, lung infection, lung cancer, etc.) over the past 10 years in China.
  2. to explore the trend of the causes of hospitalization of respiratory tumor patients (pulmonary embolism, airway stenosis, post-surgical complications, lung infection, pneumothorax, tuberculosis, etc.) in China over the past 10 years.
  3. to explore the trend of the proportion of each tumor in the respiratory department (brain tumor, nasopharyngeal cancer, thyroid cancer, lung cancer, breast cancer, liver cancer, etc.) over the past 10 years in China.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaohong Xie, Study Chair — The First Affiliated Hospital of Guangzhou Medical University
Locations (1):
- Chengzhi Zhou, Guangdong, Guangzhou, China